CLINICAL TRIAL: NCT06353217
Title: Pilot Study of a Primary Care Hypoglycemia Prevention Program
Brief Title: Study of a Primary Care Hypoglycemia Prevention Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00419034; K23DK128572 (NIH)
Record Dates: First submitted 2024-04-02; First posted 2024-04-09 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Pre/post pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient Involvement (Other): Patients who participate in the study will undergo one Baseline Clinic Visit (baseline usual care), and one Intervention clinic visit.
  Interventions: Other: Patient Group (Hypoglycemia Prevention Program)
- Primary Care Physician (PCP) Involvement (Other): PCPs will be given access to the Hypoglycemia Prevention toolkit
  Interventions: Other: Primary Care Physician Group
- Clinic Staff Involvement (Other)
  Interventions: Other: Clinic Staff Group

INTERVENTIONS:
Other: Patient Group (Hypoglycemia Prevention Program) — The Hypoglycemia Prevention Program:
  The patient hypoglycemia profile - this is a set of survey questions about hypoglycemia and related aspects of diabetes care. The questions will be administered as an Epic MyChart message sent to the patient in the week prior to the clinic visit, and in the clinic waiting room on a tablet immediately prior to the patient's primary care provider visit.
  Arms: Patient Involvement
Other: Primary Care Physician Group — The provider hypoglycemia toolkit - this is the report from the patient hypoglycemia profile, which triggers a set of hypoglycemia prevention tools and patient education materials as appropriate. Primary Care Providers will not be exposed to the intervention until all of their patients have completed the Baseline Clinic Visit.
  Arms: Primary Care Physician (PCP) Involvement
Other: Clinic Staff Group — Clinic staff will provide the tablet to the participant immediately prior to the patient's primary care provider visit.
  Arms: Clinic Staff Involvement

SUMMARY:
This is a single site, pre-post pilot study. The objective is to evaluate the acceptability and feasibility of a primary care hypoglycemia prevention program for patients taking hypoglycemia-causing medications. The study will also evaluate relevant process outcomes and clinical outcomes for refining the intervention and planning for a larger efficacy trial.

ELIGIBILITY:
Inclusion criteria for patients:

* Age 18 years or older
* Diabetes mellitus by electronic health record review
* Treatment with any of the following medication classes: insulin, sulfonylureas, meglitinides
* Community dwelling (not residing in long-term care or a skilled nursing facility)
* Receiving primary care from a participating primary care provider at Johns Hopkins Internal Medicine at Green Spring Station
* The patient's primary care provider approves their participation

Exclusion criteria for patients:

* Significant cognitive impairment or dementia
* Receiving hospice or end of life care
* Any other serious illness or condition not compatible with participation as determined by the investigators
* Planning to leave area prior to end of study
* Investigator discretion

Exclusion Criteria for continuous glucose monitoring (not required for study participation):

* History of allergic skin reaction to adhesive
* Implantable pacemaker

Inclusion criteria for primary care providers:

* Practicing at Johns Hopkins Internal Medicine Green Spring Station

Exclusion criteria for primary care providers:

* Planning to leave their position prior to end of study
* Not serving as primary care provider for any included patient

Inclusion criteria for clinic staff:

* Participating in check-in at Johns Hopkins Internal Medicine Green Spring Station

Exclusion criteria for clinic staff

* Planning to leave their position prior to end of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Overall acceptability to patients | Immediately after the intervention
  Mean score for overall acceptability on patient intervention evaluation survey (developed for this study, range 1-completely unacceptable, to 5-completely acceptable)
Overall acceptability to primary care providers | Immediately after the intervention
  Mean score for overall acceptability on primary care provider intervention evaluation survey (developed for this study, range 1-completely unacceptable, to 5-completely acceptable)
Overall acceptability to clinic staff | Immediately after the intervention
  Mean score for overall acceptability on clinic staff intervention evaluation survey (developed for this study, range 1-completely unacceptable, to 5-completely acceptable)

OTHER OUTCOMES:
Intervention coherence (patients) | Immediately after the intervention
  Mean score for intervention coherence on patient intervention evaluation survey (developed for this study, range 1-strongly disagree, to 5-strongly agree)
Opportunity costs (patients) | Immediately after the intervention
  Mean score for opportunity costs on patient intervention evaluation survey (developed for this study, range 1-strongly disagree, to 5-strongly agree)
Ethicality (patients) | Immediately after the intervention
  Mean score for ethicality on patient intervention evaluation survey (developed for this study, range 1-very unfair, to 5-very fair)
Affective attitude (patients) | Immediately after the intervention
  Mean score for affective attitude on patient intervention evaluation survey (developed for this study, range 1-very uncomfortable, to 5-very comfortable)
Burden (patients) | Immediately after the intervention
  Mean score for burden on patient intervention evaluation survey (developed for this study, range 1-no effort at all, to 5-huge effort)
Self-efficacy (patients) | Immediately after the intervention
  Mean score for self-efficacy on patient intervention evaluation survey (developed for this study, range 1-very un-confident, to 5-very confident)
Perceived effectiveness (primary care providers) | Immediately after the intervention
  Mean score for perceived effectiveness on primary care provider intervention evaluation survey (developed for this study, range 1-strongly disagree, to 5-strongly agree)
Intervention coherence (primary care providers) | Immediately after the intervention
  Mean score for intervention coherence on primary care provider intervention evaluation survey (developed for this study, range 1-strongly disagree, to 5-strongly agree)
Opportunity costs (primary care providers) | Immediately after the intervention
  Mean score for opportunity costs on primary care provider intervention evaluation survey (developed for this study, range 1-strongly disagree, to 5-strongly agree)
Affective attitude (primary care providers) | Immediately after the intervention
  Mean score for affective attitude on primary care provider intervention evaluation survey (developed for this study, range 1-very uncomfortable, to 5-very comfortable)
Burden (primary care providers) | Immediately after the intervention
  Mean score for burden on primary care provider intervention evaluation survey (developed for this study, range 1-no effort at all, to 5-huge effort)
Self-efficacy (primary care providers) | Immediately after the intervention
  Mean score for self-efficacy on primary care provider intervention evaluation survey (developed for this study, range 1-Very unconfident, to 5-very confident)
Burden (clinic staff) | Immediately after the intervention
  Mean score for burden on clinic staff intervention evaluation survey (developed for this study, range 1-no effort at all, to 5-huge effort)
Opportunity costs (clinic staff) | Immediately after the intervention
  Mean score for opportunity costs on clinic staff intervention evaluation survey (developed for this study, range 1-strongly disagree, to 5-strongly agree)
Recruitment rate | Immediately after the intervention
  % of eligible participants who consented to participate
Retention rate for second clinic visit | Immediately after the intervention
  % of participants who completed two clinic visits
Continuous glucose monitoring (CGM) completion | Immediately after the final CGM measurement (4-12 weeks after the intervention)
  % of participants who completed CGM measurements
Continuous glucose monitoring (CGM) wear time | Immediately after the final CGM measurement (4-12 weeks after the intervention)
  Mean days with complete CGM data
Time needed to complete patient hypoglycemia profile | Immediately after completion of intervention clinic visit
  Mean completion time (minutes) for patient hypoglycemia profile
Duration of clinical visit | Change from baseline to immediately after completion of intervention clinic visit
  Change from baseline in mean duration of clinic visit (minutes)
Patient completion of hypoglycemia assessment | Immediately after completion of intervention clinic visit
  Completion rate overall and for individual items
Primary care provider use of provider hypoglycemia toolkit | Immediately after completion of intervention clinic visit
  Rate of toolkit use overall and for individual tools
Patient hypoglycemia burden on continuous glucose monitoring (CGM) | Baseline to post-intervention up to 12 weeks
  Change from baseline in mean minutes per day with glucose <70 mg/dl and <54 mg/dl
Patient time below range on continuous glucose monitoring (CGM) | Baseline to post-intervention up to 12 weeks
  Change from baseline in % time with glucose <70 mg/dl
Patient time above range on continuous glucose monitoring (CGM) | Baseline to post-intervention up to 12 weeks
  Change from baseline in % time with glucose >180 mg/dl
Patient mean glucose on continuous glucose monitoring (CGM) | Baseline to post-intervention up to 12 weeks
  Change from baseline in mean glucose
Patient satisfaction with care | Change from baseline to immediately after the intervention
  Change from baseline in mean score on The Patient Satisfaction Questionnaire Short Form (PSQ-18), range 1 (lowest satisfaction) to 5 (highest satisfaction) in 7 domains
Patient activation | Change from baseline to immediately after the intervention
  Change from baseline in mean score on Patient Activation Measure (PAM 10), range 0 (lowest activation) to 100 (highest activation)
Patient self-reported hypoglycemic events | Change from baseline to 4-12 weeks after the intervention
  Change from baseline in frequency of level 1, level 2, and level 3 hypoglycemia events on hypoglycemia history survey
Changes to hypoglycemia-causing medications | Change from baseline to immediately after the intervention
  % of patients with changes in diabetes medications (dose increase, decrease, stop, switch, initiate)
Glucagon prescription | Change from baseline to immediately after the intervention
  % of patients with active glucagon prescription
Continuous glucose monitoring (CGM) prescription | Change from baseline to immediately after the intervention
  Change from baseline in frequency of CGM prescription
Change in Frequency of Referrals to Diabetes Self Management Training (DSMT) | Change from baseline to immediately after the intervention
  Change from baseline in frequency of DSMT referral
Frequency of hypoglycemia history discussions | Change from baseline to immediately after the intervention
  Frequency and content of hypoglycemia history discussion by audio-recording
Frequency of Hypoglycemia anticipatory guidance discussions | Change from baseline to immediately after the intervention
  Frequency, content, and accuracy of hypoglycemia anticipatory guidance
Frequency of Medication adherence discussions | Change from baseline to immediately after the intervention
  Frequency and content of discussions of adherence to diabetes medications

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Pilla, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States